CLINICAL TRIAL: NCT05454644
Title: Effectiveness of a Person-centred Prescription Model in Hospitalised Geriatric Patients at the End of Life
Brief Title: Effectiveness of a Person-centred Prescription Model at the End of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matia Foundation (Other)
Collaborators: University of the Basque Country (UPV/EHU) (Other); Universidad de León (Other)
Responsible Party: Principal Investigator, Alexander Ferro Uriguen, Dr, Matia Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PCP-EOL
Record Dates: First submitted 2022-06-30; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: End-Of-Life; Inappropriate Prescribing; Deprescriptions; Palliative Medicine; Geriatrics
MeSH Terms: conditions — Death

STUDY DESIGN:
Intervention Model Description: Comparison of person-centred prescription model application versus standard pharmaceutical care alone. The intervention is applied randomly during hospital stay in hospitalised older people at the end of life. The primary outcome is the mean change between admission and discharge in the number of regular medications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Pharmaceutical Care (No Intervention): Patients in the control arm receive usual pharmaceutical care in hospital. Reconciliation of the medication at hospital admission and a validation of the treatment modifications during the hospitalisation is carried out.
- Person-Centred Prescription Model (Experimental): An interdisciplinary medicine-optimisation strategy is implemented in people at the end of life (EOL) based on the person-centred prescription (PCP).
  Interventions: Other: Person-Centred Prescription Model

INTERVENTIONS:
Other: Person-Centred Prescription Model — Step 1: Identify patients with advanced chronic condition and limited life expectancy.
  Step 2: Interview with patients or closes caregiver.
  Step 3: Medication Review
  The clinical pharmacist conduct a structured medication review based on the medication appropriateness index (MAI):
  * Indication/effectiveness: Product information, STOPPFrail (Screening Tool of Older Persons' Prescriptions in Frail adults with limited life expectancy) criteria and Beers Criteria for Potentially Inappropriate Medication Use in Older Adults.
  * Dosage adjustment: Product Information and Lexi-Comp's Geriatric Dosage Handbook.
  * Correct and practical directions: Medication Regimen Complexity Index (MRCI).
  * Drug-drug interactions: Bot Plus/Beers Criteria and drug burden index (DBI), which measures dose-dependent anticholinergic and sedative loads.
  * Drug-disease interactions: Beers Criteria.
  * Duplication, duration and cost-effectiveness: Product information.
  Step 4: Treatment Plan
  Arms: Person-Centred Prescription Model

SUMMARY:
This study's main objective is to investigate whether the application of an adapted person-centred prescription model during a hospital stay would reduce the use of inappropriate or futile regular medications in older people at the end of life, improving their clinical/health statuses and reducing the expense associated with pharmacological treatment. We hypothesised that applying this modified method could optimise pharmacotherapeutic indicators and the expense associated with the pharmacological treatment of hospitalised patients

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the geriatric convalescence unit and identified as having a non-oncological advanced chronic disease and being in need of palliative care, with a limited survival prognosis according to the necessity of palliative care (NECPAL) test.

Exclusion Criteria:

* Patients with hospital stays of less than 72 hours.
* Patients transferred to other hospitals or units.
* Patients with imminently terminal patients.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Change between admission and discharge in the number of regular medications. | 3 months

SECONDARY OUTCOMES:
Change between admission and discharge in the STOPP Frail Criteria | 3 months
Change between admission and discharge in the Drug Burden Index (DBI) | 3 months
Change between admission and discharge in the total drug-drug interactions | 3 months
Change between admission and discharge in the Medication Regimen Complexity Index (MRCI) | 3 months
Change in the 28-day cost of prescriptions in € | 3 months
Number of patients who have had a new emergency department presentation. | 3 months
Number of patients who have had unplanned hospital readmission | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Matia Foundation, Donostia / San Sebastian, Gipuzkoa, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Mahony D, O'Connor MN. Pharmacotherapy at the end-of-life. Age Ageing. 2011 Jul;40(4):419-22. doi: 10.1093/ageing/afr059. Epub 2011 May 28. PMID 21622981
- [Background] Espaulella-Panicot J, Molist-Brunet N, Sevilla-Sanchez D, Gonzalez-Bueno J, Amblas-Novellas J, Sola-Bonada N, Codina-Jane C. [Patient-centred prescription model to improve adequate prescription and therapeutic adherence in patients with multiple disorders]. Rev Esp Geriatr Gerontol. 2017 Sep-Oct;52(5):278-281. doi: 10.1016/j.regg.2017.03.002. Epub 2017 May 2. Spanish. PMID 28476211
- [Background] Thompson W, Lundby C, Graabaek T, Nielsen DS, Ryg J, Sondergaard J, Pottegard A. Tools for Deprescribing in Frail Older Persons and Those with Limited Life Expectancy: A Systematic Review. J Am Geriatr Soc. 2019 Jan;67(1):172-180. doi: 10.1111/jgs.15616. Epub 2018 Oct 13. PMID 30315745
- [Background] Hanlon JT, Schmader KE, Samsa GP, Weinberger M, Uttech KM, Lewis IK, Cohen HJ, Feussner JR. A method for assessing drug therapy appropriateness. J Clin Epidemiol. 1992 Oct;45(10):1045-51. doi: 10.1016/0895-4356(92)90144-c. PMID 1474400
- [Background] Lavan AH, Gallagher P, Parsons C, O'Mahony D. STOPPFrail (Screening Tool of Older Persons Prescriptions in Frail adults with limited life expectancy): consensus validation. Age Ageing. 2017 Jul 1;46(4):600-607. doi: 10.1093/ageing/afx005. PMID 28119312
- [Background] By the American Geriatrics Society 2015 Beers Criteria Update Expert Panel. American Geriatrics Society 2015 Updated Beers Criteria for Potentially Inappropriate Medication Use in Older Adults. J Am Geriatr Soc. 2015 Nov;63(11):2227-46. doi: 10.1111/jgs.13702. Epub 2015 Oct 8. PMID 26446832
- [Background] George J, Phun YT, Bailey MJ, Kong DC, Stewart K. Development and validation of the medication regimen complexity index. Ann Pharmacother. 2004 Sep;38(9):1369-76. doi: 10.1345/aph.1D479. Epub 2004 Jul 20. PMID 15266038
- [Background] Hilmer SN, Mager DE, Simonsick EM, Cao Y, Ling SM, Windham BG, Harris TB, Hanlon JT, Rubin SM, Shorr RI, Bauer DC, Abernethy DR. A drug burden index to define the functional burden of medications in older people. Arch Intern Med. 2007 Apr 23;167(8):781-7. doi: 10.1001/archinte.167.8.781. PMID 17452540
- [Background] Potter K, Flicker L, Page A, Etherton-Beer C. Deprescribing in Frail Older People: A Randomised Controlled Trial. PLoS One. 2016 Mar 4;11(3):e0149984. doi: 10.1371/journal.pone.0149984. eCollection 2016. PMID 26942907
- [Derived] Ferro-Uriguen A, Beobide-Telleria I, Gil-Goikouria J, Pena-Labour PT, Diaz-Vila A, Herasme-Grullon AT, Echevarria-Orella E, Seco-Calvo J. Application of a person-centered prescription model improves pharmacotherapeutic indicators and reduces costs associated with pharmacological treatment in hospitalized older patients at the end of life. Front Public Health. 2022 Oct 3;10:994819. doi: 10.3389/fpubh.2022.994819. eCollection 2022. PMID 36262221